CLINICAL TRIAL: NCT00198952
Title: Effects of Herbal Products on Metabolism and Hunger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Natural Prescriptions (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NP2000-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2002-04

CONDITIONS: Obesity; Metabolism
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Drug: DietPro
Drug: Placebo

SUMMARY:
to test safety and efficacy on metabolism, heart rate, blood pressure, TSH (and other blood)and hunger/caloric compensation on ephedra versus placebo

ELIGIBILITY:
Inclusion Criteria:

age 18-50, non-smoking, not pregnant (serum), Beck <15, physician permission

Exclusion Criteria:

pregnant, lactating, smoker, use of appetite-affecting medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2000-02; Study Completion 2001-03

PRIMARY OUTCOMES:
metabolic rate
heart rate
blood pressure
TSH
caloric compensation

SECONDARY OUTCOMES:
weight
body composition

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States